CLINICAL TRIAL: NCT06932224
Title: Hospital-associated Deconditioning: Exploring Factors Contributing to the Physical and Cognitive Decline of Older Adults During Hospitalisation
Brief Title: This Study Aims to Measure the Effect of Acute Hospitalisation on the Physical and Cognitive Functioning of Older Orthopaedic Patients (Aged 65 or Above).
Status: Recruiting | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: RHM MED2068
Record Dates: First submitted 2025-03-26; First posted 2025-04-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-12

CONDITIONS: Deconditioning; Orthopedic Fractures; Hospital Associated Deconditioning; Orthopaedic Injuries
Keywords: Hospital acquired deconditioning; Hospital associated deconditioning; Physical functioning; Cognitive functioning; Orthopaedic; Older patient; Older adults (65 years and older); Muscle strength; Muscle mass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Older patients with orthopaedic conditions/injuries: This cohort will take part in the physical and cognitive questionnaires and tests at all 3 (4 if interim is needed) time points.
  20 patients of this cohort will take part in one semi-structured interview.
- Southampton General Hospital Staff: 10 hospital staff to take part in one semi-structured interview.

SUMMARY:
This study aims to investigate the impact of hospitalisation on physical and cognitive performance in patients aged 65 and older admitted with an orthopaedic injury. This will be achieved by asking patients to participate in a series of physical and cognitive performance questionnaires and tests. These questionnaires and tests will be performed by the patients as close to their admission as possible and then again at day 7 of hospitalisation (or discharge if earlier) and at 4-6 weeks after discharge. However, if a patient's hospital stay lasts more than 30 days, they will be asked to take part in the interim data collection timepoint.

To summarize, patients will be assessed at least 3 times, 4 if your hospital stay is longer than 30 days. The first and second assessments will be in the hospital, and the third will be 4-6 weeks after discharge at you home (or where is appropriate). Additionally, patients will be asked to wear an activity watch between the first and second assessment.

The study will also explore patients experiences of their hospital stay and opinions on deconditioning, including the views and opinions of hospital staff. This information will be gathered by having interviews with a sample of the patients who took part in the questionnaires and tests and by having interviews with hospital staff. The interview will be conducted by the main researcher, Thomas Cartledge, and will take place either over the phone, online or in-person, depending on your preference. The interviews will be audio and/or video recorded, however the recordings will be deleted immediately once transcription is completed. The duration of the interview will last approximately 30-60 mins.

ELIGIBILITY:
Patient criteria:

Inclusion:

* Older adults aged 65 years or older
* Able to provide written consent
* Admitted to Southampton General Hospital (SGH) for an acute orthopaedic condition
* Been admitted to SGH <72 hours before recruitment

Exclusion:

* Older adults who are not able to safely complete the quantitative measurement tools, as advised by the patient's clinician
* Patients receiving end of life care
* Require a hoist to transfer from bed to chair prior to hospitalisation
* Been admitted to SGH >72 hours before recruitment
* Unable to consent

Hospital staff criteria:

Inclusion:

* Work at SGH
* Work with older orthopaedic inpatients
* Be able to provide written consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults admitted to SGH with an acute orthopaedic condition/injury.
  Hospital staff who work at SGH who work with older orthopaedic inpatients.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Muscle strength measured via a hand held dynamometer. | From enrolment to the last data collection point at 4-6 weeks post discharge
Muscle mass measured via Bioelectrical Impedance Analysis. | From enrolment to the last data collection point at 4-6 weeks post discharge.
  The specific measure used will be fat free mass (FFM)
Sarcopenia risk assessed via the SARC-F questionnaire. | From enrolment to the last data collection point at 4-6 weeks post discharge.
  Strength, assistance with walking, rising from a chair, climbing stairs, and falls (SARC-F) questionnaire.
  Using a scale ranging from 0 to 10, with a higher score indicating a higher sarcopenia risk.
Functional mobility measured via the Short Physical Performance Battery (SPPB) questionnaire. | 4-6 weeks (discharge to the final data collection point).
  The SPPB score ranges from 0 to 12 points, with a higher score indicating better functional mobility.
Health-related quality of life measured by the EQ-5D questionnaire. | From enrolment to the last data collection point at 4-6 weeks post discharge.
  The EuroQol-5D (EQ-5D) is a two part questionnaire. The first part is a descriptive system using five dimensions to describe health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression).
  The second part is a visual analogue scale (VAS) where participants indicate their overall health by drawing a line on a scale from 100 (best imaginable health) to 0 (worst imaginable health).
Physical function measured via the Barthel Index questionnaire. | From enrolment to the last data collection point at 4-6 weeks post discharge.
  The original Barthel Index will be used, which uses a score ranging from 0 to 100. A higher score indicates a better physical function.
Cognitive impairment measured via The Montreal Cognitive Assessment (MoCA) score. | From enrolment to the last data collection point at 4-6 weeks post discharge.
  The MoCA score ranges from 0 to 30. A score of 26 or higher is generally considered normal, with lower scores indicating potential cognitive impairment.
Delirium measured via the 4AT score. | From enrolment to the last data collection point at 4-6 weeks post discharge.
  The 4AT test is scored from 0-12. A score of 0 suggests no delirium and no moderate-severe cognitive impairment. A score from 1-3 suggests cognitive impairment but not delirium. A score of 4 or more suggest delirium.

SECONDARY OUTCOMES:
Hospital re-admission rate | 3 months
  Will see if patients are readmitted to hospital within 3 months. Information abstracted from medical records.
Hospital re-admission rate | 6 months
  Will see if patients are readmitted to hospital within 6 months. Information abstracted from medical records.

OTHER OUTCOMES:
Perceptions and attitudes towards hospital-associated deconditioning measured via semi-structured interviews. | Time frame for patients will be their last hospital admission (approx 7 days long) and staff will be asked to recall information from their last 2 months of work.
  Interviews will be conducted with older orthopaedic patients and hospital staff.
Exploring practical ways of preventing hospital-associated deconditioning via semi-structed interviews. | Time frame for patients will be their last hospital admission (approx 7 days long) and staff will be asked to recall information from their last 2 months of work.
  Interviews will be conducted with older orthopaedic patients and hospital staff.
Exploring barriers and facilitators to physical and cognitive risk factors of hospital-associated deconditioning via semi-structed interviews. | Time frame for patients will be their last hospital admission (approx 7 days long) and staff will be asked to recall information from their last 2 months of work.
  Interviews will be conducted with older orthopaedic patients and hospital staff.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Southampton Foundation Trust, Southampton, Hampshire, United Kingdom